CLINICAL TRIAL: NCT07374081
Title: Autism Spectrum Disorder and Criminal Responsibility in the Italian Forensic Context - Multicenter Study for Italian Validation of the Forensic Autism Risk Assessment Scale.
Brief Title: Italian Validation of the Forensic Autism Risk Assessment Scale (FARAS-IT)
Acronym: ASD_FARASIT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Felice Carabellese, FULL PROFESSOR, University of Bari
Other Study IDs: ASD FARAS-IT
Record Dates: First submitted 2026-01-05; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder (ASD
Keywords: ASD,; FARAS,; Italian Criminal Justice,; Forensic Psychiatry; SPJ
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Perpetrators in Forensic Psychiatric context: Group A comprises all perpetrators of criminal offenses who, during the observation period, are subject to psychiatric security measures, both detentive (for example, REMS) and non-detentive (such as probation with therapeutic prescriptions)
- Perpetrators considered criminally responsible: Group B includes subjects who are perpetrators of criminal offenses that do not result in being managed as psychiatric patients
- Psychiatric patients' non-perpetrators of offenses: Group C comprises psychiatric patients who have never committed offenses, followed by territorial mental health services

SUMMARY:
The study is a multicenter observational project designed to translate, culturally adapt, and validate the Italian version of the FARAS (FARAS-IT), a structured framework for assessing risk and protective factors specific to individuals with Autism Spectrum Disorder (ASD) involved in the Italian criminal justice system.

Adult participants (≥18 years) with a diagnosis or well-founded clinical suspicion of ASD are consecutively enrolled over 12 months into three groups: offenders in forensic psychiatric settings under security measures, offenders considered criminally responsible and not under psychiatric care, and psychiatric patients with ASD without any history of criminal behavior followed by community mental health services or non-forensic residential facilities.

All participants undergo assessment with FARAS-IT and complementary clinical and forensic instruments (e.g., WHODAS 2.0, BPRS or equivalents, HCR-20, SAPROF, DUNDRUM), alongside collection of clinical, functional, and judicial variables, in order to evaluate the psychometric properties of FARAS-IT (factor structure, internal consistency, test-retest and inter-rater reliability, convergent and discriminant validity) and its clinical-forensic usefulness in understanding criminal responsibility and judicial decision-making trajectories in individuals with ASD.

DETAILED DESCRIPTION:
The study is a multicenter, observational project aimed at translating, culturally adapting, and validating the Forensic Autism Risk Assessment Scale (FARAS-IT) for use in the Italian criminal responsibility context. It focuses on adults with Autism Spectrum Disorder (ASD) or well-founded clinical suspicion of ASD who are involved in different forensic and clinical settings, with the overarching goal of improving the structured assessment of vulnerability, risk, and protective factors relevant to criminal responsibility and judicial decision-making.

The research is designed as a non-randomized, cross-sectional, comparative cohort study with prospective enrollment of all eligible participants over a 12-month observation period (T0), with standardized data collection at the time of clinical-forensic or clinical evaluation. Participants are recruited in three Italian regions (Campania, Apulia, and Tuscany) from a range of contexts that reflect different degrees of involvement with the criminal justice and mental health systems, ensuring a heterogeneous and representative sample.

Three groups are included: Group A consists of perpetrators of criminal offenses managed in forensic psychiatric pathways and subject to detentive or non-detentive security measures (e.g., REMS, forensic residential and intermediate facilities, probation with therapeutic prescriptions); Group B includes perpetrators of offenses who are considered criminally responsible and are managed in correctional facilities or external criminal execution settings without a psychiatric treatment pathway; Group C comprises psychiatric patients with ASD who have never committed criminally relevant acts and are followed in community mental health services or non-forensic residential or semi-residential facilities. This tripartite structure allows the study to distinguish between factors associated with ASD per se and those specifically related to criminal behavior and forensic management.

The primary objective is to assess the psychometric properties of FARAS-IT, including internal consistency, reliability, convergent and discriminant validity, and its clinical-forensic utility across these settings. Secondary objectives include: clinically and forensically characterizing adults with ASD in different judicial and health contexts; exploring the associations between FARAS profiles, indicators of criminal responsibility, expert findings, and judicial outcomes; identifying under-diagnosed ASD among perpetrators not in psychiatric care; and evaluating the incremental contribution of FARAS-IT beyond traditional risk and functioning instruments such as HCR-20, SAPROF, DUNDRUM, and WHODAS 2.0.

FARAS-IT is administered to subjects with a diagnosis or well-founded suspicion of ASD and covers seven domains of autistic functioning that are particularly relevant for forensic formulations (e.g., social communication, cognitive rigidity, cognitive empathy, adaptability, sensory sensitivity, emotional regulation, and risk awareness). Data are gathered through clinical interviews, behavioral observation, and analysis of clinical and, where available, forensic documentation, and are integrated-when applicable-into existing forensic information systems such as the SMOP registry for patients in forensic psychiatric circuits.

All participants provide written informed consent, with specific attention to the vulnerability of forensic and correctional populations and to the communicative and cognitive characteristics associated with ASD. Consent procedures and information delivery are adapted using clear, concrete language, sufficient time for explanation, and, when needed, simplified communication supports; in cases of reduced decision-making capacity, legal guardians or administrators are involved in accordance with Italian law, while always seeking the participant's assent.

Data are pseudonymized and managed in line with EU Regulation 2016/679 (GDPR) and national legislation, with identifying information stored separately from clinical and psychometric datasets and accessible only to authorized personnel. Statistical analyses follow current psychometric and forensic psychiatry standards (e.g., COSMIN recommendations) and include descriptive analyses, exploratory and confirmatory factor analyses, reliability estimates, and comparative models to test the discriminatory capacity of FARAS-IT among the three groups and its relationship with judicial and clinical outcomes.

Ultimately, the study aims to provide the first systematic Italian validation of FARAS in a large, clinically and forensically diverse ASD population, contributing to more structured, transparent, and reproducible evaluations of criminal responsibility and procedural competence in individuals on the autism spectrum.

ELIGIBILITY:
Inclusion Criteria: Subjects will be included in the study who meet all of the following criteria:

* age 18 years or older;
* diagnosis of Autism Spectrum Disorder formally made according to DSM-5-TR criteria or well-founded clinical suspicion of ASD, documented by specialist evaluation;
* insertion in one of the contexts provided for groups A, B, or C;
* capacity to provide valid informed consent, clinically assessed, or presence of guardian/administrator of substance in cases provided by current law;
* sufficient language and cognitive competence to participate in the evaluation, including with autism-informed communicative adaptations.

The inclusion criterion based on *well-founded clinical suspicion* is consistent with the study's objective of intercepting the phenomenon of ASD under-diagnosis in adulthood, particularly in forensic and correctional contexts.

-

Exclusion Criteria: Subjects presenting one or more of the following conditions will be excluded from the study:

* acute medical conditions or clinical instability preventing participation in the evaluation;
* acute psychotic state, severe disorganization of thought, or substance intoxication not stabilized at the time of assessment (with possibility of subsequent re-evaluation);
* severe intellectual disability or cognitive compromise making any structured data collection impossible, even with adaptive supports;
* refusal of informed consent. Exclusion will not be based on the type of offense, in order to avoid selective bias in the sample composition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Apulia, Campania and Tuscany
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
FARAS-IT total score | Baseline (T0), at enrollment
  Total score on the Italian version of the Forensic Autism Risk Assessment Scale (FARAS-IT), calculated as the sum of item ratings across seven domains (social communication, cognitive rigidity, cognitive empathy, adaptability, sensory sensitivity, emotional regulation, risk awareness). Higher total scores indicate greater autism-related vulnerability in the forensic context.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carabellese, F., & Felthous, A. R. (2016). Forensic psychiatric evaluation and criminal responsibility. *International Journal of Law and Psychiatry*, 49, 83-90.
- [Background] Romano, M. (2018). *Imputabilità e responsabilità penale*. Milano: Giuffrè.
- [Background] Fiandaca, G., & Musco, E. (2020). *Diritto penale. Parte generale*. Bologna: Zanichelli.
- [Background] Mantovani, F. (2019). *Diritto penale. Parte generale*. Padova: CEDAM.